CLINICAL TRIAL: NCT00434538
Title: A Multicenter, Prospective, Randomized Comparison Study of BST-DERMON Versus Standard of Care in the Treatment of Diabetic Foot Ulcers
Brief Title: BST-DERMON Versus Standard of Care in the Treatment of Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to Sponsor's financial reasons
Sponsor: BioSyntech Canada Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DO-CIP01-P
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic; Foot; Ulcer; Neuropathic; Chitosan
MeSH Terms: conditions — Diabetic Foot; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BST-DermOn

SUMMARY:
This trial is designed to investigate the therapeutic benefits of using BST-DermOn for the wound repair of diabetic neuropathic foot ulcers.

The objective of this study is to evaluate the safety and efficacy of BST-DermOn in providing a clinically significant advantage over the standard of care in the repair of diabetic foot ulcers.

DETAILED DESCRIPTION:
This trial is designed to investigate the therapeutic benefits of using BST-DermOn for the wound repair of diabetic neuropathic foot ulcers. BST-DermOn is a sterile, non-toxic, nonpyrogenic wound dressing composed of an aqueous mixture of Chitosan, hydrochloric acid (HCl) and disodium beta-glycerol phosphate (β-GP) designed to address current wound healing needs. Chitosan has well documented wound healing properties as well as inherent haemostatic and bacteriostatic capabilities. BST-DermOn is used in conjunction with a defined standard of care and is applied over a prepared and debrided ulcer and covered with a semi-occlusive secondary dressing.

This prospective, multi-center, randomized, controlled study will enrol 130 type 1 or type 2 diabetic subjects presenting with a Grade 1 or Grade 2 (Wagner classification) diabetic foot ulcer of 1-10cm² on the mid or forefoot. Subjects who meet the eligibility criteria will be assigned to one of two groups:

1. a control group that will receive the standard of care or
2. a treatment group that will receive BST-DermOn.

Treatments in both groups will be applied three (3) times a week for up to twenty consecutive weeks or until the study ulcer is closed. All subjects will be followed for safety and efficacy during treatment visits through a final evaluation visit. There will be a post treatment follow-up visit at 4 weeks post-closure for subjects with complete re-epithelialization.

The objective of this study is to evaluate the safety and efficacy of BST-DermOn in providing a clinically significant advantage over the standard of care in the repair of diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Between eighteen (18) and eighty (80) years of age
* Type 1 or Type 2 diabetes mellitus
* Diabetes is under adequate control
* Diabetic foot ulcer located on the mid or forefoot
* Diabetic foot ulcer has been present for at least four (4) weeks and no more than two (2) years prior to screening
* Diabetic foot ulcer is ≥ 1.0cm² and ≤10cm² in size
* Diabetic foot ulcer is grade 1 or 2 according to the Wagner Grading system.

Exclusion Criteria:

* Ulcer is over an active Charcot deformity of the mid-foot ("Rocker-Bottom Foot") or over the talus, distal calcaneous, navicular, or cuboid bones or a deformity that interfere with off-loading in the opinion of the investigator
* Ulcer due to a non-diabetic aetiology
* Ulcer has tunnels or sinus tracts that cannot be completely debrided.
* Clinical evidence of infection
* Osteomyelitis
* Subject has vasculitis, severe rheumatoid arthritis, other collagen or vascular diseases or other medical conditions, outside of diabetes, known to impair wound healing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with closed ulcers at week 12

SECONDARY OUTCOMES:
Reduction in size of the diabetic foot ulcer at week 20.
Safety by analysis of AEs.
Reduction of incidence of clinical signs of infection.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Restrepo, M.D., Study Director — Medical Monitor, BioSyntech Canada Inc
Locations (20):
- Canada (20):
  - Foothills Medical Center Col Belcher Hospital, Calgary, Alberta
  - Surrey Memorial Hospital Fraser Health Authority, Surrey, British Columbia
  - Infection Control Unit, Infectious Diseases and Medical Microbiology, University of Manitoba Health Sciences Centre, Winnipeg, Manitoba
  - Dermadvance Research, Winnipeg, Manitoba
  - James Paton Memorial Hospital, Gander, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Riverside Professional Centre, Sydney River, Nova Scotia
  - The Mayer Institute, Hamilton, Ontario
  - Wassay Gezhig Na Nahn Dah We Igamig, Kenora, Ontario
  - Parkwood Hospital, London, Ontario
  - Dermatology Clinic, Mississauga, Ontario
  - EntraLogix Clinical Group, Newmarket, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Dermatology Daycare and Wound Healing Clinic, Toronto, Ontario
  - Centre podiatrique, Boucherville, Quebec
  - Clinique de dermatologie Giard & Toscano, 500 Greber #110, Gatineau, Quebec
  - Centre de Recherche Clinique de Laval, Laval, Quebec
  - CHAU-Hôtel-Dieu de Lévis, Département de médecine de jour- 5ème étage, Clinique des plaies complexes, Lévis, Quebec
  - CHUM - Hotel Dieu, Montreal, Quebec
  - St-Jerome Medical Research Inc., Saint-Jérôme, Quebec

REFERENCES:
- See also: Sponsor website — http://www.biosyntech.com